CLINICAL TRIAL: NCT03110159
Title: Cyclic PDT for the Prevention of Actinic Keratosis and Non Melanoma Skin Cancer in Solid Organ Transplant Recipients
Brief Title: DUSA: Cyclic PDT for the Prevention of AK & NMSC in Solid Organ Transplant Recipients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Medical Dermatology Specialists (Other)
Collaborators: DUSA Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PHXB-16-0142-80-15; MDS (Other: Medical Dermatology Specialists)
Record Dates: First submitted 2017-03-15; First posted 2017-04-12 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Skin Cancer; Non-melanoma Skin Cancer; Sun Damaged Skin; Actinic Keratosis
Keywords: Photodynamic therapy; Prevention; Actinic Keratosis; Skin Cancer; Non-melanoma Skin Cancer; Sun Damaged Skin; Solid Organ Transplant; PDT
MeSH Terms: conditions — Skin Neoplasms; Keratosis, Actinic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Levulan® Kerastick® and blue light illumination (Experimental): Levulan® Kerastick® for Topical Solution will be applied to a designated area for 3 hours without occlusion prior to illumination with blue light using the standard FDA approved treatment time for the BLU-U device of 16 minutes 40 seconds.
  Each subject will be randomized to undergo treatment to one side face and one dorsal forearm/hand treatment, while the other side will serve as untreated control. Treatments will be conducted at the beginning of study Day 1 (Initial Treatment), Day 30 after the initial treatment (+ 3 days), Day 180 after initial treatment (+ 30 days), 1 year after the initial treatment (+ 30 days), and every 6 months (+ 30 days) thereafter for 2 additional years.
  Interventions: Drug: Levulan® Kerastick®; Drug: BLU-U Blue Light Photodynamic Therapy

INTERVENTIONS:
Drug: Levulan® Kerastick® — Levulan® Kerastick® for Topical Solution will be applied to a designated area for 3 hours without occlusion prior to illumination with blue light
Drug: BLU-U Blue Light Photodynamic Therapy — 3 hours after Levulan® Kerastick® for Topical Solution is applied blue light illumination of designated area will be performed using the standard FDA approved treatment time of 16 minutes 40 seconds.
  Other Names: blue light illumination

SUMMARY:
This is a pilot, phase 2, prospective, comparative study to evaluate the safety and efficacy of the combination of Levulan® Kerastick® for Topical Solution and blue light illumination using the BLU-U® Blue Light Photodynamic Therapy Illuminator (LevulanPDT).

The study hypothesis is that post solid organ transplantation patients, highly susceptible to non-melanoma skin cancer, can be treated safely and effectively through clinical cyclic application of PDT, lessening morbidity and possible mortality for this immunosuppressed patient population.

ELIGIBILITY:
Inclusion Criteria:

* Received solid organ transplant
* 3-24 months post-transplant (any number of transplant)
* Time interval of at least 6 days duration where complications such as rejection episodes, viral infections, surgical interventions and therapies with mono or polyclonal antibodies are ruled out by the transplant team.
* No prior history of NMSC in the treatment fields
* No AK/Bowen's disease in the treatment fields within the last 3 months.
* Moderate to severe sun damage
* Be willing to forego other interventions in the treatment fields than the ones approved by the investigator that would interfere with the protocol or evaluation of the study medication

Exclusion Criteria:

* Patients with Fitzpatrick's scale skin type IV-VI
* Cutaneous photosensitivity to wavelengths of 400-450 nm, porphyria or known allergies to porphyrins
* Known sensitivity to any of the components of the Levulan® Kerastick® for Topical Solution
* Prior use of topical or systemic therapies that might interfere with the evaluation of the study medication during the study, within a 3 month washout period from the time of the screening visit
* Unable to return for follow-up visits and tests
* Any condition or situation which in the Investigator's opinion may put the subject at significant risk, could confound the study results, or could interfere significantly with the subject's participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-08-29 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
Primary prevention of AKs in recently transplanted solid organ recipient | 3 Years
  Number of AK will be counted for each site using the photographs of the treatment and the control areas. AKs will be graded by thickness.
Time to occurrence of AKs in recently transplanted solid organ recipient | 3 Years
  Time to occurrence of AK will be calculated from the first visit to the development of an AK in the treatment areas and in the control areas.
Primary prevention of NMSC in recently transplanted solid organ recipient | 3 Years
  Number of NMSC will be counted for each site using the photographs of the treatment and the control areas. NMSC, including basal cell carcinoma, Bowen's disease and squamous cell carcinoma, will be diagnosis and confirmed histologically by biopsy.
Time to occurrence of NMSC in recently transplanted solid organ recipient | 3 Years
  Time to occurrence of NMSC will be calculated from the first visit to the development of an NMSC in the treatment areas and in the control areas.

SECONDARY OUTCOMES:
Pain control with Levulan-PDT in Solid Organ Transplant Recipient | Day 1, Day 30, Day 180, 12 months, 18 months, 24 months, 30 months, 36 months
  Pain will be assessed on the 10 point Visual Analogue Scale (VAS), as mild (0-3), moderate (4-7) or severe (8-10). Patients will be asked to rate the pain at the beginning, midway point (approximately 8 minutes later), and at the end of each PDT session.
The number of participants with treatment related adverse events as assessed by the CTCAE v4.0 | 3 Years
  The number of evaluable study participants who had a grade 3 or higher adverse event (AE) or any serious adverse event that's determined to be at least possibly or probably related to study treatment, or any AE which is at least possibly or probably related to study treatment that causes permanent study discontinuation.

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie C. Zeitouni, MD, Principal Investigator — Medical Dermatology Specialists
Locations (1):
- Medical Dermatology Specialists, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-06): https://cdn.clinicaltrials.gov/large-docs/59/NCT03110159/Prot_SAP_000.pdf